CLINICAL TRIAL: NCT05424419
Title: Retrospektive Analyse Der Konservativen Skoliosetherapie - Doppelkorsettversorgung Mittels Tag- Und Nachtorthese Versus Ganztagesorthese
Brief Title: Add-on Nighttime Bracing in Adolescent Idiopathic Scoliosis
Status: Completed | Type: Observational
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Sponsor
Other Study IDs: EK 27012018
Record Dates: First submitted 2022-06-15; First posted 2022-06-21 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Scoliosis
Keywords: scoliosis; nighttime bracing; full-time bracing; Chêneau brace; Charleston brace
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- double-brace group: AIS patients with daytime and nighttime braces
  Interventions: Procedure: Brace therapy
- single-brace group: AIS patients with a single brace for day and night
  Interventions: Procedure: Brace therapy

INTERVENTIONS:
Procedure: Brace therapy — A Chêneau-type brace was made to be worn as a full-time brace or during daytime only (double-brace group), whereas the nighttime brace was produced according to the Charleston approach.

SUMMARY:
Bracing is an accepted standard therapy for idiopathic scoliosis at Cobb angle ranges between 25° and 45°. However, it is unclear, if a specifically tailored regimen of daytime and nighttime braces (=double brace) yields superior results compared to the standard treatment (single brace for day and night). These two treatment regimens were investigated in the study.

DETAILED DESCRIPTION:
One-hundred-fifteen patients with adolescent idiopathic scoliosis (AIS) were assessed before initiation of bracing treatment and at the final follow-up 2 years after deposition of the brace. They were divided into two groups: double-brace group and single-brace group. Each patient underwent clinical and radiological examinations and Cobb angles were measured.

ELIGIBILITY:
Inclusion Criteria:

* AIS
* age between 10 and 15 years (y)
* Risser's sign of 0-2
* Cobb curvature angle of 25-40°
* no previous treatment
* compliance (at least 23 h wearing time)

Exclusion Criteria:

* non-idiopathic scoliosis
* Cobb curvature angle >40°
* <10 years and >15 years for initial treatment

Ages: 10 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients with AIS were managed as recommended by SOSORT Consensus statement. Inclusion criteria were according to the Scoliosis Research Society criteria. Initial diagnostics included a clinical examination, standardized X-ray of the entire spine in standing position. Patients for whom cost coverage of double-brace therapy was denied by the health insurance company received a single full-day and nighttime Chêneau type brace treatment. All other patients received a Chêneau brace for daytime and a Charleston type nighttime bending brace. Patients who were prescribed the brace were instructed to wear it for 23 hours/day. Patients were seen at 6-month intervals, at which times we collected radiographic, clinical, orthotic, and self-reported data.
Sampling Method: Non-Probability Sample
Enrollment: 115 (Actual)
Dates: Start 1997-01-02 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
primary correction | At study inclusion with initiation of brace therapy
  Primary correction (%) of brace therapy (Cobb angle measurement)

SECONDARY OUTCOMES:
Cobb angle reduction | 2 years after deposition of the brace
  Follow-up Cobb angle (degree) in relation to the initial Cobb angle

IPD SHARING:
Plan to Share IPD: No